CLINICAL TRIAL: NCT03596827
Title: The Protective Immune Response to Attenuated Enterotoxigenic Escherichia Coli Infection in Healthy Human Subjects: A Pilot Study
Brief Title: The Protective Immune Response to Attenuated Enterotoxigenic Escherichia Coli Infection
Acronym: MIRRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NL66039.028.18
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Diarrhea
Keywords: Diarrhea; Gastroenteritis; Bacterial Infections; Escherichia Coli Infections; E.coli
MeSH Terms: conditions — Diarrhea; Gastroenteritis; Bacterial Infections; Escherichia coli Infections

STUDY DESIGN:
Intervention Model Description: The MIRRE pilot study is a randomized, double-blind dose-response, parallel human infection study in 30 healthy adults
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1E10 CFU Escherichia coli (E. coli) (Active Comparator): At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 1E10 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A dose 1E10 CFU
- 1E9 CFU Escherichia coli (E. coli) (Experimental): At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 1E9 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A dose 1E9 CFU
- 1E8 CFU Escherichia coli (E. coli) (Experimental): At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 1E8 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A dose 1E8 CFU
- 1E7 CFU Escherichia coli (E. coli) (Experimental): At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 1E7 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A dose 1E7 CFU
- 1E6 CFU Escherichia coli (E. coli) (Experimental): At day 14, after a standardized evening meal and overnight fast, subjects receive a single oral dose of 1E6 CFU of the attenuated diarrhoeagenic E. coli strain E1392-75-2A. At day 35, after a standardized evening meal and overnight fast, all subjects receive a second inoculation 1E10 CFU of the diarrhoeagenic E. coli.
  Interventions: Biological: E. coli strain E1392-75-2A dose 1E6 CFU

INTERVENTIONS:
Biological: E. coli strain E1392-75-2A dose 1E10 CFU — Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonization Factor Antigen II (CFA/II) and provides 75% protection against challenge with an LT, ST, CFA/II strain
  Arms: 1E10 CFU Escherichia coli (E. coli)
Biological: E. coli strain E1392-75-2A dose 1E9 CFU — Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonization Factor Antigen II (CFA/II) and provides 75% protection against challenge with an LT, ST, CFA/II strain
  Arms: 1E9 CFU Escherichia coli (E. coli)
Biological: E. coli strain E1392-75-2A dose 1E8 CFU — Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonization Factor Antigen II (CFA/II) and provides 75% protection against challenge with an LT, ST, CFA/II strain
  Arms: 1E8 CFU Escherichia coli (E. coli)
Biological: E. coli strain E1392-75-2A dose 1E7 CFU — Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonizat
  Arms: 1E7 CFU Escherichia coli (E. coli)
Biological: E. coli strain E1392-75-2A dose 1E6 CFU — Diarrhoeagenic E. coli strain E1392/75-2A serotype O6:H16 belongs to Pathogen class 2 . The strain has a deletion of genes encoding the heat-labile (LT) and heat-stable (ST) toxins and can not produce any toxins. However, it continues to express Colonizat
  Arms: 1E6 CFU Escherichia coli (E. coli)

SUMMARY:
The existing diarrhoeagenic Escherichia coli (E. coli) challenge model is already suitable for dietary interventions in its current form, targeted to impact on the immediate clinical symptoms upon E. coli infection. In order to make the model also suitable for dietary interventions that are aimed at support of the protective response against reinfection, the immune response triggered by the primary infection should be suboptimal. The MIRRE pilot study is set up to determine how much the primary inoculation dose of diarrheagenic E. coli should be lowered in order to result in a reduced protective response upon a secondary infection.

DETAILED DESCRIPTION:
The MIRRE pilot study is a randomized, double-blind dose-response, parallel 7 weeks human infection study. Healthy male subjects, 18-55 years of age who fulfil all of the inclusion criteria and none of the exclusion criteria, will be randomly assigned to one of five inoculation dosages of a live attenuated diarrheagenic E. coli strain (n=6 per group). Subjects will be instructed to maintain their usual pattern of physical activity and their habitual food intake, but to reduce and standardize their dietary calcium intake. After a standardized evening meal and an overnight fast, subjects will be orally infected on day 14 and 35 with a live, but attenuated, diarrheagenic E. coli (strain E1392/75-2A; collection NIZO food research). Five groups of 6 subjects will be provided one of the following dosages at day 14: 1E10 CFU (standard dose); 1E9 CFU; 1E8 CFU; 1E7 CFU or 1E6 CFU of the E.coli strain. At study day 35, all subjects will receive a second inoculation of 1E10 CFU of the E.coli strain.

At various time points before and after diarrheagenic E. coli challenges an online diary will be kept to record information on stool consistency, frequency and severity of symptoms, and blood and stool samples are collected to quantify antibody levels and to quantify fecal infection parameters.

The hypothesis of this pilot study is that the E. coli infection dose at primary inoculation determines the outcomes of the protective immune response and the extent of clinical symptoms at a secondary inoculation.Therefore the CFA/II-specific IgG antibody response, in relation to clinical symptoms, is the main outcome.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Male
2. Age between 18 and 55 years.
3. BMI ≥18.5 and ≤30.0 kg/m2.
4. Healthy as assessed by the NIZO health questionnaire.
5. Ability to follow Dutch verbal and written instructions.
6. Availability of internet connection.
7. Signed informed consent.
8. Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned.
9. Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for at least 15 years.
10. Willing to comply with study procedures, including collection of stool and blood samples.
11. Willingness to abstain from high calcium containing products.
12. Willingness to abstain from alcoholic beverages three days before, during and for 4 days after diarrheagenic E. coli challenge.
13. Willingness to abstain from medications that contain acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs, (OTC) antacids and antimotility agents (eg, loperamide) on the three days before, during and for 4 days after diarrheagenic E. coli challenge.
14. Willingness to abstain from probiotics and prebiotic/fibers starting from runin and during the whole study.
15. Willingness to give up blood donation starting at run-in and during the entire study.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Acute gastroenteritis in the 2 months prior to inclusion
2. Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus infection (HIV).
3. Disease of the GI tract, liver, gall bladder, kidney, thyroid gland (self-reported), except for appendicitis.
4. History of microbiologically confirmed ETEC or cholera infection within 3 years prior to inclusion.
5. Symptoms consistent with Travelers' Diarrhea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to inclusion, OR planned travel to endemic countries during the length of the study.
6. Vaccination for, or ingestion of cholera within 3 years prior to inclusion, including studies at NIZO.
7. Occupation involving handling of ETEC or Vibrio cholerae currently, or within 3 years prior to inclusion.
8. Vaccination for, or ingestion of ETEC or E coli heat labile toxin, including E. coli challenge studies at NIZO.
9. Evidence of current excessive alcohol consumption (>4 consumptions/day or >20 consumptions/week) or drug (ab)use, and not willing/able to stop this during the study.
10. Known allergy to the following antibiotics: ciprofloxacin, trimethoprim, sulfamethoxazole, and penicillins.
11. Reported average stool frequency of >3 per day or <1 per 2 days.
12. Use of antibiotics, (during 6 months prior to inclusion), norit, laxatives, cholestyramine, antacids H2 receptor antagonists or proton pump inhibitors (during 3 months prior to inclusion).
13. Use of immunosuppressive drugs (e.g. cyclosporine, azathioprine, systemic corticosteroids, antibodies).
14. Vegans.
15. Mental status that is incompatible with the proper conduct of the study.
16. Not having a general practitioner, not allowing disclosure of participation to the general practitioner or not allowing to inform the general practitioner about abnormal results.
17. Participation in any clinical trial including blood sampling and/or administration of substances starting 1 month prior to study start and during the entire study.
18. Personnel that is part of the study team at NIZO, their partner and their first and second degree relatives.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity is self-reported by the subjects through a questionnaire.
Enrollment: 30 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in specific antibody titer | Day 14,21,28 and Day 35,42,49
  Serum IgG-CFA/II antibody levels in relation to clinical symptoms at second E.coli inoculation

SECONDARY OUTCOMES:
Change in percentage of faecal wet weight from baseline | Day 11,12 and Day 15-17. Day 33,34 and 36-38
  % of faecal wet weight determined by freeze-drying
Change in Stool consistency (Bristol stool scale) from baseline | Day 11-17 and Day 32-38
  Stool consistency for all stools reported by the subjects
Change in Stool frequency from baseline | Day 11-17 and Day 32-38
  Stools per day reported by the subjects
Change in incidence, duration and severity of Gastro-intestinal symptoms from baseline | Day 11-17 and Day 32-38
  Gastro-intestinal Symptom Rating Scale reported by the subjects in the online diary

CONTACTS AND LOCATIONS:
Overall Officials: Melle van Schaik, Study Director — NIZO Food Research
Locations (1):
- NIZO Food Research, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bovee-Oudenhoven IM, Lettink-Wissink ML, Van Doesburg W, Witteman BJ, Van Der Meer R. Diarrhea caused by enterotoxigenic Escherichia coli infection of humans is inhibited by dietary calcium. Gastroenterology. 2003 Aug;125(2):469-76. doi: 10.1016/s0016-5085(03)00884-9. PMID 12891550
- [Background] Ten Bruggencate SJ, Girard SA, Floris-Vollenbroek EG, Bhardwaj R, Tompkins TA. The effect of a multi-strain probiotic on the resistance toward Escherichia coli challenge in a randomized, placebo-controlled, double-blind intervention study. Eur J Clin Nutr. 2015 Mar;69(3):385-91. doi: 10.1038/ejcn.2014.238. Epub 2014 Nov 5. PMID 25369827
- See also: Sponsor information — http://www.nizo.com